CLINICAL TRIAL: NCT00031902
Title: Rituxumab Combined With Chemotherapy (PVB) For Poor Prognosis HIV-Related Non-Hodgkin's Lymphoma
Brief Title: Rituximab Plus Combination Chemotherapy in Treating Patients With HIV-Related Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lymphoma Trials Office (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069238; BNLI-POORRISKHIV; EU-20145
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2003-02

CONDITIONS: Lymphoma
Keywords: AIDS-related peripheral/systemic lymphoma; AIDS-related diffuse large cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related small noncleaved cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma; AIDS-related lymphoblastic lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Bleomycin; Rituximab; Prednisolone; Vincristine

INTERVENTIONS:
Biological: bleomycin sulfate
Biological: rituximab
Drug: prednisolone
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Monoclonal antibodies such as rituximab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining rituximab with chemotherapy may kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of rituximab plus combination chemotherapy in treating patients who have HIV-related non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with poor-prognosis, HIV-related non-Hodgkin's lymphoma treated with rituximab combined with prednisolone, vincristine, and bleomycin.
* Determine the toxicity of this regimen in these patients.
* Determine the time to progression and survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive chemotherapy comprising vincristine IV and bleomycin IV on day 1 and oral prednisolone every other day beginning on day 1. Treatment repeats every 3 weeks for 6 courses. Patients also receive rituximab on days 14, 21, 28, and 35. Patients who achieve complete response (CR) receive 2 additional courses of chemotherapy after CR.

Patients are followed every 1-2 months.

PROJECTED ACCRUAL: A total of 10-20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of poor-prognosis, HIV-related non-Hodgkin's lymphoma (HIV-NHL)

  * Previously untreated
* More than 1 of the following criteria:

  * Prior diagnosis of AIDS
  * ECOG performance status 3-4
  * CD4 count less than 100/mm3
* No primary cerebral lymphoma

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* See Disease Characteristics

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for HIV-NHL
* At least 1 year since prior chemotherapy for Kaposi's sarcoma (KS)

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior radiotherapy for HIV-NHL allowed
* At least 1 year since prior radiotherapy for KS

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-10

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Pettengell, MD, Study Chair — St. George's Hospital
Locations (2):
- United Kingdom (2):
  - St. George's Hospital, London, England
  - Chelsea Westminster Hospital, London